CLINICAL TRIAL: NCT05508490
Title: Prevalence of Acute Kidney Injury in Patients With Diabetic Ketoacidosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Refaat Fathy, resident doctor, Assiut University
Other Study IDs: AKI in DKA
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: AKI in Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: renal chemistry, serum electrolyte, — detection of renal chemistry affection and electrolyte disturbance in diabetic ketoacidosis

SUMMARY:
prevalence of acute kidney injury in patients with diabetic ketoacidosis

DETAILED DESCRIPTION:
Acute kidney injury (formerly known as acute renal failure) is a syndrome characterised by the rapid loss of the kidney's excretory function and is typically diagnosed by the accumulation of end products of nitrogen metabolism (urea and creatinine) or decreased urine output, or both.

* Stages of kidney injury:

  1. Risk: 1.5 folds increase in serum creatinine and urine output less than 0.5 ml/kg/hr for 6 hours.
  2. Injury: two folds increase in serum creatinine and urine output less than 0.5 ml/kg/hr for 12 hours.
  3. Failure: three folds increase in serum creatinine and urine output less than 0.3 ml/kg/hr for 24 hours or anuria for 12 hours.
  4. Loss: complete loss of kidney function > 4 weeks
  5. End stage kidney disease: complete loss of kidney function > 3 months It is the clinical manifestation of several disorders that affect the kidney acutely. Acute kidney injury is common in hospital patients and very common in critically ill patients. In these patients, it is most often secondary to extrarenal events. How such events cause acute kidney injury is controversial. No specific therapies have emerged that can attenuate acute kidney injury or expedite recovery; thus, treatment is supportive. New diagnostic techniques (eg, renal biomarkers) might help with early diagnosis. Patients are given renal replacement therapy if acute kidney injury is severe and biochemical or volume-related, or if uraemic-toxaemia-related complications are of concern. If patients survive their illness and do not have premorbid chronic kidney disease, they typically recover to dialysis independence. However, evidence suggests that patients who have had acute kidney injury are at increased risk of subsequent chronic kidney disease.

     Children with diabetic ketoacidosis (DKA) are at significant risk for various degrees of dehydration and disruption of electrolyte balance due to osmotic diuresis [1]. As a consequence of chronic polyuria, progressive dehydration is common in patients with DKA [2]. Children are less likely to establish the compensatory process for dehydration than adults, making them more vulnerable to dehydration [3]. In patients with extreme volume loss, pre-renal acute kidney injury (AKI) is likely, and acute tubular necrosis can occur. As the rate of glomerular filtration decreases, there is insufficient kidney acid excretion, thereby aggravating metabolic acidosis [4]. Since metabolic acidosis normalization is one of the goals of DKA management [1], AKI can adversely affect recovery from metabolic acidosis for these patients. Besides, AKI is an independent risk factor for a prolonged hospital stay and increased mortality rates [5]. DKA is managed by volume resuscitation, insulin therapy, and correction of electrolyte imbalances [6]. Resuscitation using traditional saline in DKA patients can exacerbate electrolyte abnormalities, in particular the production of hyperchloremia [7, 8]. While an increase of evidence suggests that hyperchloremia is linked to an increased risk of morbidity and mortality, its effects in DKA are not well defined [9, 10].

     Aim of study 1: to detect prevalence of acute kidney injury in pediatric patients with diabetic ketoacidosis and its impact as regard to;
* duration of hospital stay.
* Occurance of complications
* response to treatment. 2: to detect the type of kidney injury in diabetic ketoacidosis wether it is renal or pre renl.

Type of study Observational Cross-Sectional study

Sample size Sample size will be determined through statistical analysis by Public health department

Patients and methods All included children were subjected to

1. detailed medical history including demographic data (name, age, and sex), age of onset, family history of type 1 diabetes mellitus (DM1), and duration of the disease, previous attacks of DKA.
2. clinical examination with particular emphasis on assessment of anthropometric measures (weight and height), evaluation of systolic and diastolic blood pressures, monitoring of urine output (UOP), and recording of complications (cerebral edema, sepsis, need for vasoactive drugs, need for respiratory support and mortality).
3. laboratory investigations including daily urine output, urea, creatinine, serum chloride level, Na, K and arterial blood gases (ABG) every third day and albumin/creatinine ratio (ACR) every week.

Follow-up of blood urea and creatinine till normalization of kidney function or occurance of failure.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion was children with DKA with an age range between 1 and 18 years

Exclusion Criteria:

* The exclusion criteria were patients with septic shock, acute pancreatitis, and chronic kidney disease and patients who received fluid therapy before referral to our hospital

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All included children were subjected to
  1. detailed medical history including demographic data (name, age, and sex), age of onset, family history of type 1 diabetes mellitus (DM1), and duration of the disease, previous attacks of DKA.
  2. clinical examination with particular emphasis on assessment of anthropometric measures (weight and height), evaluation of systolic and diastolic blood pressures, monitoring of urine output (UOP), and recording of complications (cerebral edema, sepsis, need for vasoactive drugs, need for respiratory support and mortality).
  3. laboratory investigations including daily urine output, urea, creatinine, serum chloride level, Na, K and arterial blood gases (ABG) every third day and albumin/creatinine ratio (ACR) every week.
  Follow-up of blood urea and creatinine till normalization of kidney function or occurance of failure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of acute kidney injury in diabetic ketoacidosis | Baseline
  detection of renal function affection and electrolyte disturbance in patients with diabetic ketoacidosis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang EM, Lee HG, Oh KY, Kim CJ. Acute Kidney Injury in Pediatric Diabetic Ketoacidosis. Indian J Pediatr. 2021 Jun;88(6):568-573. doi: 10.1007/s12098-020-03549-9. Epub 2020 Nov 19. PMID 33210207